CLINICAL TRIAL: NCT06111599
Title: Thermovision-controlled Lumbar Sympathetic Blockade in Chronic Limb-threatening Ischemia Treatment
Acronym: Tevi-LuSy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Europainclinics z.ú. (Other)
Collaborators: Slovak Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4/2023/VUSCH/EK
Record Dates: First submitted 2023-10-21; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Chronic Limb-Threatening Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Patients with chronic limb-threatening ischemia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Proximal arterial obliteration
  Interventions: Procedure: lumbar sympathetic blockade
- Group B (Experimental): Distal arterial obliteration
  Interventions: Procedure: lumbar sympathetic blockade
- Group C (Experimental): Complex arterial obliteration
  Interventions: Procedure: lumbar sympathetic blockade

INTERVENTIONS:
Procedure: lumbar sympathetic blockade — Skiascopic-guided lumbar sympathetic blockade with the administration of local anesthetic

SUMMARY:
Thermovision-controlled lumbar sympathetic blockade in chronic limb-threatening ischemia treatment

DETAILED DESCRIPTION:
Chronic limb-threatening ischemia (CLTI), the end-stage of lower extremity artery disease (LEAD), occurs with growing prevalence around the globe and is associated with increased healthcare costs. CLTI is defined by the presence of LEAD in combination with rest pain, gangrene, or lower limb ulceration lasting more than two weeks. Despite unclear results of abdominal surgical lumbar sympathectomy, novel interventional minimally invasive fluoroscopy-guided procedures seem to be promising. A prospective interventional study will be conducted, primarily targeting patients afflicted by critical limb ischemia, with the incorporation of thermal vision control and tissue oxygen monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Chronic limb-threatening ischemia-Patients with chronic leg pain for at least 6 months with intensity (VAS >=5)
* those who (only if a signature was obtainable), or whose legal guardian,fully understood the clinical trial -details and signed the informed consent form

Exclusion Criteria:

* Chronic Venous Insufficiency
* women with positive a pregnancy tests before the trial or who planned to become pregnant within the following 3 years
* other patients viewed as inappropriate by the staff
* disagreement with participation in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-22 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline EuroQoL-5 Dimension (EQ-5D) Value 3m | 3 months follow-up
  EQ-5D-5L self-care, usual activities, pain/discomfort and anxiety/depression
Change From Baseline EuroQoL-5 Dimension (EQ-5D) Value 6m | 6 months follow-up
  EQ-5D-5L self-care, usual activities, pain/discomfort and anxiety/depression
Change From Baseline Visual Analog Pain Scale (VAS) of Back Pain 3m | 3 months follow-up
  Change From Baseline Visual Analog Pain Scale (VAS) of Back Pain 3m measured by VAS 10 point measurement
Change From Baseline Visual Analog Pain Scale (VAS) of Back Pain 6m | 6 months follow-up
  Change From Baseline Visual Analog Pain Scale (VAS) of Back Pain 6m measured by VAS 10 point measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Europainclinics, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided
numerical rating scale of quality of life

REFERENCES:
- [Derived] Kocan L, Rajtukova V, Rasiova M, Kocanova H, Hudak R, Vaskova J, Satnik V, Martuliak I, Hudak M. Infrared monitoring-based optimization of interventional lumbar sympathectomy outcomes evaluation in peripheral vascular disease patients: Experimental trial thermovision-guided lumbar sympathectomy. Medicine (Baltimore). 2025 Feb 14;104(7):e41524. doi: 10.1097/MD.0000000000041524. PMID 39960937